CLINICAL TRIAL: NCT04767594
Title: PERFORM: An EPidEmiological, PRospective Cohort Study to Generate Real-world Evidence in Patients With HR+/HER2- Advanced Breast Cancer Treated in the First Line Setting as Per Current Standard Of Care With an EndocRine-based Palbociclib CoMbination Therapy
Brief Title: First-line Palbociclib and Endocrine Therapy for Patients With HR+/HER2- Advanced Breast Cancer in the Real-world Setting.
Acronym: PERFORM
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481152; PERFORM-NIS (Other: Alias Study Number)
Record Dates: First submitted 2021-01-21; First posted 2021-02-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First-line Palbociclib + endocrine therapy: Palbociclib + letrozole, or Palbociclib + anastrozole, or Palbociclib + exemestane, or Palbociclib + fulvestrant after prior endocrine therapy
  Interventions: Drug: Palbociclib + endocrine therapy

INTERVENTIONS:
Drug: Palbociclib + endocrine therapy — Palbociclib + letrozole, or Palbociclib + anastrozole, or Palbociclib + exemestane, or Palbociclib + fulvestrant after prior endocrine therapy In pre- or perimenopausal women, the endocrine therapy should be combined with a luteinizing hormone-releasing hormone (LHRH) agonist.

SUMMARY:
This is a prospective, single-arm, multi-center observational non-interventional study (NIS) in Germany and Austria.

DETAILED DESCRIPTION:
Patients diagnosed with HR+/HER2- locally advanced or metastatic breast cancer indicated by their treating physicians for first line endocrine-based palbociclib combination therapy and who meet eligibility criteria will be invited to participate in this study. The key objectives of this study are to describe clinical, scientific and patient reported outcomes for patients with HR+/HER2- locally advanced or metastatic breast cancer initiating treatment with first line endocrine-based palbociclib combination therapy in the real-world setting in Germany and Austria. Patient characteristics, real-world treatment patterns, treatment sequences and reasons for the physician's treatment decisions will be collected. Additional real-world research questions are to explore patient-focused parameters such as longitudinal follow-up data on patient-reported outcomes beyond disease progression and by treatment sequence or to analyze the time from the start of first line treatment to the first administered palliative chemotherapy. Clinical outcome by treatment sequences will be described. Routinely assessed biomarkers and diagnostic procedures applied for treatment sequence decisions will be collected.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
2. Diagnosis of HR+/HER2- locally advanced, inoperable or metastatic breast cancer.
3. Physician has determined that first-line treatment with palbociclib (i) in combination with an aromatase inhibitor, or (ii) in combination with fulvestrant in women who received prior endocrine therapy as per current local product label is indicated. In pre- or perimenopausal women, the endocrine therapy should be combined with a luteinizing hormone-releasing hormone (LHRH) agonist.
4. Patients who in the opinion of the investigator are willing and able to comply with regular clinic visits as per local standard of care practice at the study site.
5. Age of 18 years or older.

Patients meeting any of the following criteria will not be included in the study:

1. Any contraindication as per current local product label.
2. Prior systemic antineoplastic treatment for advanced disease. Exception: Start of first line treatment with palbociclib in combination with aromatase inhibitor or fulvestrant as per current local product label is allowed up to 4 weeks prior to inclusion.
3. Patients currently participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. Note: A concomitant participation in other non-interventional/observational studies, registries and translational research networks (e.g., PRAEGNANT, OPAL) or chart reviews is allowed.
4. Patients who are unable to understand the nature of the study or are unwilling to sign an informed consent.

Patient eligibility should be reviewed, documented, and confirmed by an appropriately qualified member of the investigator's study team before patients are enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HR+/HER2- locally advanced or metastatic breast cancer indicated by their treating physicians for first line endocrine-based palbociclib combination therapy and who meet eligibility criteria will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1409 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | from date of start of first-line treatment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 7.5 years

SECONDARY OUTCOMES:
Cohort-specific PFS of second-line treatment | from date of start of second-line treatment until the date of first subsequent documented disease progression or date of death from any cause, whichever came first, assessed up to 7.5 years
  Cohorts are defined by substance class of second-line therapy following first-line endocrine-based palbociclib therapy
Cohort-specific PFS2 | from date of start of first-line treatment until the date of documented disease progression on the respective second-line treatment or date of death from any cause, whichever came first, assessed up to 7.5 years
Landmark progression-free survival rates (PFSR) of first- and second-line treatment | proportion of patients without documented disease progression or death due to any cause at defined intervals after start of first-/second-line treatment (at 6, 12, 18, 24, 30, 36 months)
Overall survival (OS) | from date of start of first-line treatment until the date of documented death from any cause, assessed up to 7.5 years
Landmark overall survival rates (OSR) | proportion of patients without documented death due to any cause at defined intervals (at 12, 24, 36, 48, 60 months after start of first-line treatment)
Objective response rate (ORR) of first- and second-line treatment | from date of start of first-/ second-line treatment until the date of first subsequent documented disease progression or date of death from any cause, whichever came first, assessed up to 7.5 years
Duration of response (DoR) of first- and second-line treatment | from the date of first documented tumor response during first-/ second-line treatment until to the date of first subsequent documented disease progression or to death due to any cause, whichever came first, assessed up to 7.5 years
Disease control rate (DCR) of first- and second-line treatment | proportion of patients with documented tumor response during first-/second-line treatment (as assessed by local investigator in routine clinical practice) or stable disease (SD) over a period of at least 24 weeks after start of first-line treatment
Progression-free survival (PFS) of third-line treatment | from date of start of third-line treatment until the date of first subsequent documented disease progression or date of death from any cause, whichever came first, assessed up to 7.5 years
Time to first subsequent therapy (TFST) | from date of start of first-line treatment until the date of start of first subsequent systemic antineoplastic treatment, assessed up to 7.5 years
Time to first subsequent chemotherapy (TFSC) | from date of start of first-line treatment until the date of start of first subsequent systemic chemotherapy or chemotherapy-based antineoplastic treatment, assessed up to 7.5 years
Change from baseline in the FACT-B total score | from the date of first questionnaire assessment until the date of last questionnaire assessment, assessed at baseline, thereafter 3-monthly until end of study, and at the end of palbociclib treatment, up to 7.5 years.
  The FACT-B is a 37-item instrument designed to measure five domains of Health-Related Quality of Life (HRQOL) in breast cancer patients: Physical Well-being (PWB), Social/family Well-being (SWB), Emotional Well-being (EWB), Functional Well-being (FWB) as well as a Breast Cancer Subscale (BCS).
  Utilized with the 27 core FACT-G items, the FACT-B was developed with an emphasis on patients' values and brevity.
  For all questions, participants are asked to respond to a 5-point Likert-type scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The higher the score, the better the QOL (minimum 0; maximum 148).
Change from baseline in the FACT-G total score | from the date of first questionnaire assessment until the date of last questionnaire assessment, assessed at baseline, thereafter 3-monthly until end of study, and at the end of palbociclib treatment, up to 7.5 years.
  The FACT-G is a 27-item instrument designed to measure four domains of HRQOL in breast cancer patients: PWB, SWB, EWB, and FWB.
  For all questions, participants are asked to respond to a 5-point Likert-type scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The higher the score, the better the QOL (minimum 0; maximum 108).
Change from baseline in the FACT-B subscales scores: PWB, SWB, EWB, FWB and additional concerns for BCS. | from the date of first questionnaire assessment until the date of last questionnaire assessment, assessed at baseline, thereafter 3-monthly until end of study, and at the end of palbociclib treatment, up to 7.5 years.
  The FACT-B is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients: PWB, SWB, EWB, FWB as well as a BCS. Utilized with the 27 core FACT-G items, the FACT-B was developed with an emphasis on patients' values and brevity.
  For all questions, participants are asked to respond to a 5-point Likert-type scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The higher the score, the better the QOL (PWB: minimum 0; maximum 28. SWB: minimum 0; maximum 28. EWB: minimum 0; maximum 24. FWB: minimum 0; maximum 28. BCS: minimum 0; maximum 40).
Change from baseline in FACT-B Trial Outcome Index (TOI) | from the date of first questionnaire assessment until the date of last questionnaire assessment, assessed at baseline, thereafter 3-monthly until end of study, and at the end of palbociclib treatment, up to 7.5 years.
  The FACT-B is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients: PWB, SWB, EWB, FWB as well as a BCS. Utilized with the 27 core FACT-G items, the FACT-B was developed with an emphasis on patients' values and brevity. The TOI combines the PWB+FWB+BCS items, making it 24-items altogether.
  For all questions, participants are asked to respond to a 5-point Likert-type scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The higher the score, the better the QOL (minimum 0; maximum 96).
Time to deterioration (TTD) in FACT-B total score | From the date of first questionnaire assessment until the date of first subsequent questionnaire with a decrease of ≥ 7 points in FACT-B total score or death, whichever came first, assessed up to 7.5 years.
  The FACT-B is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients: PWB, SWB, EWB, FWB as well as a BCS. Utilized with the 27 core FACT-G items, the FACT-B was developed with an emphasis on patients' values and brevity.
  For all questions, participants are asked to respond to a 5-point Likert-type scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The higher the score, the better the QOL (minimum 0; maximum 148).
Landmark analyses of cohort-specific Area Under the Curve (AUC) in the Functional Assessment of Cancer Therapy - Breast (FACT-B) TOI-Physical/Functional/Breast (TOI-PFB) | From the date of first questionnaire assessment until 12, 24, 36, 48 months thereafter (irrespective of disease or treatment situation at that time point)
  Cohorts are defined by substance class of second-line therapy following first-line endocrine-based palbociclib therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (191):
- Austria (9):
  - Sankt Josef Hospital Braunau, Braunau am Inn
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Country Hospital Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Priv. Doz. OA Dr. Michael Hubalek, Schwaz
  - Medizinische Universität Wien, Abteilung Innere Medizin I, Vienna
  - Medizinische Universität Wien, Vienna
  - Oesterreichische Gesundheitskasse Hanusch-Krankenhaus, Vienna
- Germany (182):
  - Klinikum Bayreuth GmbH, Bayreuth, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Medizinische Universität Lausitz Carl Thiem, Cottbus, Brandenburg
  - Onkologische Kooperation Harz, Goslar, Lower Saxony
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim, Other
  - Mvz Etgo Gmbh, Berlin, Other
  - Onkologisch-Hämatologische Schwerpunktpraxis, Bremen, Other
  - ANregiomed gKU, Ansbach
  - Alexianer Klinikum Hochsauerland GmbH, Arnsberg
  - Group practice Heinrich, Augsburg
  - Group Practice Steinfeld-Birg, Augsburg
  - Group practice Tanzer, Bad Reichenhall
  - Group practice Seipelt, Bad Soden a.T.
  - Klinikum Mittelbaden Baden-Baden Balg, Baden-Baden
  - Sozialstiftung Bamberg Klinikum am Bruderwald, Bamberg
  - Private Practice Bayreuth, Bayreuth
  - Charité Campus Mitte, Berlin
  - Hämatologie Onkologie Berlin-Mitte, Berlin
  - MediOnko-Institut GbR, Berlin
  - DRK Kliniken Berlin-Köpenick Brustzentrum, Berlin
  - Vivantes MVZ Hellersdorf - Zweigpraxis Biesdorf, Berlin
  - Group practice Morack, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Frauenarzt-Zentrum-Zehlendorf, Berlin
  - Dr. Leonid Basovski Hämatologikum Biberach, Biberach an der Riss
  - Evangelisches Klinikum Bethel gGmbH, Klinik für Innere Medizin, Hämatologie, Onkologie, Bielefeld
  - Group practice Bueckner, Bochum
  - Praxiskooperation Onkologie Bonn / Euskirchen / Rheinbach / Wesseling GbR, Bonn
  - Group practice Hannig, Bottrop
  - Marienhospital Bottrop gGmbH, Bottrop
  - ONKO DOK GbR, Bottrop
  - Kliniken Boeblingen, Böblingen
  - Staedtisches Klinikum Brandenburg GmbH, Brandenburg
  - Private practice Brandenburg a.d.H., Brandenburg a.d.H.
  - Klinikum Bremerhaven Reinkenheide gGmbH, Bremerhaven
  - Fürst-Stirum-Klinik Bruchsal Klinik für Frauenheilkunde und Geburtshilfe, Bruchsal
  - AKH-Gruppe-Allgemeines Krankenhaus Celle + MVZ gGmbH, Celle
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Private Practice Jungberg, Chemnitz
  - private practice Ziegler-Loehr, Cologne
  - St. Elisabeth Krankenhaus GmbH, Cologne
  - St. Vincenz-Krankenhaus, Datteln
  - Onkologiezentrum Donauwoerth, Donauwörth
  - Klinikum Dortmund Frauenklinik, Dortmund
  - Studiengesellschaft Gefos Dortmund mbH, Dortmund
  - Group practice Goehler, Dresden
  - Gemeinschaftspraxis, Dresden
  - Group practice Jacobasch, Dresden
  - Naedler GmbH, Duisburg
  - St. Marien-Hospital, Düren
  - Private Practice Groell, Ebersberg
  - Studienzentrale für das MVZ Eggenfelde e.K., Eggenfelden
  - St. Georg Klinikum Eisenach gGmbH, Eisenach
  - Group practice Weniger, Erfurt
  - Group practice Haecker, Erlangen
  - imland gGmbH, Fockbek
  - Universitaetsklinikum Frankfurt Frauenheilkunde, Frankfurt am Main
  - pioh Studien und Management GbR, Frechen
  - Group Practice Dr. med. M. Zaiss, Freiburg im Breisgau
  - KKH Landkreis Freudenstadt Frauenheilkunde und Geburtshilfe, Freudenstadt
  - Group practice Fuerth, Fürth
  - MVZ II der Niels Stensen Kliniken, Georgsmarienhütte
  - Onkostudien Gera GbR, Gera
  - Private practice Rabenbauer, Grafenau
  - Klinikum Oberberg KKH Gummersbach, Gummersbach
  - Onkodok GmbH, Gütersloh
  - Group practice Neumeister, Haldensleben I
  - Group practice Behlendorf, Halle
  - Studiengesellschaft Haemato-Onkologie Hamburg GbR, Hamburg
  - Praxisklinik Harburger Ring, Hamburg
  - Katholisches Marienkrankenhaus gGmbH Frauenklinik, Hamburg
  - Überörtliche Gemeinschaftspraxis, Hamburg
  - Private Practice Rubanov, Hamelin
  - Klinikum Hanau Gynäkologisches Krebszentrum, Hanau
  - Group Practice Kamal, Hanover
  - Westkuestenkliniken Heide und Brunsbuettel, Heide
  - Private Practice Fuxius, Heidelberg
  - Private practice Petersen, Heidenheim a.d.B.
  - Mathilden-Hospital, Herford
  - cancer Center Zweiseenland GbR, Herrsching am Ammersee
  - Private Practice Dr. med. Andreas Lorenz, Hildburghausen
  - Gemeinschaftspraxis Dr.med. Ch. Uleer, Hildesheim
  - Onkologie Hof MVZ GmbH, Hof
  - Universitätsklinik des Saarlandes Ausführende Stelle: Universitätsklinikum Homburg,, Homberg (Efze)
  - Frauenarzt Toralf Baerens, Ilsede
  - Klinikum Itzehoe, Itzehoe
  - IDGGQ GbR, Kaiserslautern
  - ViDia Christliche Kliniken Karlsruhe Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Diakonissenkrankenhaus Karlsruhe, Karlsruhe
  - Klinikum Kaufbeuren, Kaufbeuren
  - Institut fuer Versorgungsforschung in der Onkologie GbR, Koblenz
  - Klinikum Dahme-Spreewald GmbH, Königs Wusterhausen
  - group practice Krefeld, Krefeld
  - Private practice Kronach, Kronach
  - Klinikum Kulmbach, Kulmbach
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH Landshut, Landshut
  - Group practice Koehler, Langen
  - Onkologisches Zentrum Lebach, Lebach
  - Group practice Mueller, Leer
  - Group practice Knoblich, Loerrach
  - Private practice Wierick, Lohsa
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Onkologie Zentrum Lüneburg Praxisgemeinschaft, Lüneburg
  - Universitätsklinikum Magdeburg Frauenklinik, Brustzentrum, Magdeburg
  - Klinikum Magdeburg Frauenheilkunde und Geburtshilfe, Magdeburg
  - Group practice Prof. Dr. M. Hensel, Mannheim
  - Klinikum Fichtelgebirge gGmbH, Marktredwitz
  - Hämatologisch Onkologisches Studieninstitut, Mayen
  - MVZ Hämatologie/Onkologie, Mayen
  - OnkoLog Moers GbR, Moers
  - Brustzentrum-Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - Stauferklinikum Schwaebisch Gmuend, Mutlangen
  - MVZ GmbH-Muehlhausen, Mühlhausen
  - Onko - Log Muelheim GbR, Mühlheim
  - Klinikum Dritter Orden, München
  - Group practice Schmidt, München
  - Private practice Naunhof, Naunhof
  - Dr Ines Vanselor Gessner U A Kagelmacher, Neubrandenburg
  - Group Practice Nacke, Neuenahr-Ahrweller
  - Friedrich-Ebert-Krankenhaus, Neumünster
  - TZN-Tumorzentrum Niederrhein GmbH, Neuss
  - Spital 2 medizinisches Institut PartG mbB, Nuremberg
  - medius Klinik Nürtingen, Nürtingen
  - ONSO GbR, Oldenburg
  - Pius Hospital Oldenburg, Oldenburg
  - Oberhavel Kliniken GmbH, Oranienburg
  - Klinikum Osnabrueck GmbH, Osnabrück
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - MVZ für Hämatologie und Onkologie, Ravensburg
  - Oncologianova GmbH, Recklinghausen
  - Group practice Remscheid, Remscheid
  - Private practice Remscheid, Remscheid
  - Onkologie Zentrum Süd MVZ GmbH, Remscheid
  - Gemeinschaftspraxis für internistische Hämatologie und Onkologie, Rheine
  - Nadler GmbH, Rinteln
  - Private practice Markmann, Rostock
  - Klinikum Suedstadt Rostock, Universitaetsfrauenklinik, Rostock
  - Agaplesion Diakonieklinik Rotenburg gGmbH, Rotenburg (Wümme)
  - GPR Klinikum Rüsselsheim, Rüsselsheim am Main
  - CaritasKlinikum St. Theresia, Saarbrücken
  - Krankenhaus Saarlouis vom DRK, Saarlouis
  - Private practice Schubert, Scheibenberg
  - MedCenter Nordsachsen - Studien, Schkeuditz
  - Onkster GbR, Schorndorf
  - Diakoneo Diakonie-Klinikum Schwaebisch Hall gGmbH, Schwäbisch Hall
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH, Schweinfurt
  - Marienkrankenhaus Schwerte, Schwerte
  - Group Practice Esser, Siegburg
  - Group practice Singen, Singen (Hohentwiel)
  - Onkologiezentrum Soest/Iserlohn, Soest
  - Staedtisches Klinikum Solingen gemeinützige GmbH, Klinik für Frauenheilkunde, Solingen
  - KMG Klinikum Sömmerda, Sömmerda
  - Group practice Behringer, Speyer
  - MVZ Klinik Dr. Hancken GmbH, Stade
  - Johanniter-Krankenhaus Genthin Stendal, Stendal
  - Private Practice Denck, Stendal
  - Clinical Research Stohlberg GmbH, Stohlberg
  - Private practice Stralsund, Stralsund
  - Gynäkologie Kompetenzzentrum Praxis Dr. med. Carsten Hielscher, Stralsund
  - Klinikum der Landeshauptstadt Stuttgart gKAoeR, Stuttgart
  - Vinzenz von Paul Kliniken gGmbH Marienhospital, Stuttgart
  - Frauenaerztliches Zentrum Suhl im medico Facharztzentrum MVZ GmbH Betriebsstaette Suhl, Suhl
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Group Practice Kronawitter, Traunstein
  - Klinikum Traunstein, Traunstein
  - Group practice Forstbauer, Troisdorf
  - Private practice Weissenborn, Twistringen
  - Group practice Wagner, Völklingen
  - GRN Klinik Weinheim, Weinheim
  - Asklepios Klinik Weissenfels Frauenheilkunde, Geburtshilfe Brustzentrum, Weißenfels
  - MVZ Marien-Hospital Wesel GmbH, Wesel
  - Medizinische Studiengesellschaft NORD-WEST GmbH, Westerstede
  - Lahn-Dill-Kliniken GmbH, Wetzlar
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Gruop practice Rodemer / Wismann / Distelrath, Wilhelmshaven
  - Rems-Murr-Klinikum Winnenden Gynaekologie und Geburtshilfe, Winnenden
  - GIM - Gemeinschaftspraxis Innere Medizin, Witten
  - Group practice Wolfsburg, Wolfsburg
  - Helios Universitätsklinikum Wuppertal GmbH, Wuppertal
  - Group practice Wuerzburg, Würzburg
  - Universitätsklinikum Wuerzburg AoeR, Würzburg

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lux MP, Runkel ED, Glastetter E, Vannier C, Buncke J, Frank M, Bartsch R, Thill M, Wockel A. PERFORM: a non-interventional study assessing the patients' treatment starting with 1L palbociclib in HR+/HER2- ABC. Future Oncol. 2022 Nov;18(36):3971-3982. doi: 10.2217/fon-2022-0552. Epub 2022 Nov 25. PMID 36427183
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481152